CLINICAL TRIAL: NCT07321704
Title: Effect of Antiseptic Irrigations With 0.05% Chlorhexidine Gluconate (Irrisept) Versus Normal Saline on Fasciocutaneous Flap-Based Closure of Pilonidal Disease With Myriad Extracellular Matrix Implantation
Brief Title: Effect of Antiseptic Irrigations With 0.05% Chlorhexidine Gluconate (Irrisept) Versus Normal Saline on Fasciocutaneous Flap-Based Closure of Pilonidal Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yosef Nasseri, MD (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Sponsor-Investigator, Yosef Nasseri, MD, Principal Investigator, Nasseri,Yosef MD
Organization: Nasseri,Yosef MD (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00091579
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pilonidal Disease
MeSH Terms: interventions — Therapeutic Irrigation; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1: Irrisept (0.05% Chlorhexidine Gluconate) Irrigation (Experimental): Participants undergoing bilateral gluteal fasciocutaneous flap closure with implantation of Myriad extracellular matrix will receive intraoperative wound irrigation using Irrisept (0.05% chlorhexidine gluconate) according to the surgeon's standard technique. Irrigation is applied immediately before surgical closure.
  Interventions: Device: Irrisept (0.05% chlorhexidine gluconate)
- Arm 2: Normal Saline Irrigation (Standard of Care) (Active Comparator): Participants undergoing bilateral gluteal fasciocutaneous flap closure with implantation of Myriad extracellular matrix will receive intraoperative wound irrigation using sterile normal saline, consistent with current standard surgical practice.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Device: Irrisept (0.05% chlorhexidine gluconate) — Irrisept solution will be used to irrigate the surgical wound prior to flap closure. The solution is applied using manufacturer-recommended technique and volume. No other changes to surgical care are made.
  Other Names: Chlorhexidine gluconate wound lavage; CHG 0.05% irrigation
  Arms: Arm 1: Irrisept (0.05% Chlorhexidine Gluconate) Irrigation
Other: Normal Saline — Sterile normal saline will be used to irrigate the surgical wound prior to flap closure according to the surgeon's standard technique. No antiseptic agents will be added.
  Other Names: Sterile saline; standard irrigation
  Arms: Arm 2: Normal Saline Irrigation (Standard of Care)

SUMMARY:
Pilonidal disease is a chronic condition that causes painful inflammation and infection near the top of the buttocks. Many patients require surgery, and one commonly used approach is a bilateral gluteal fasciocutaneous flap with midline closure along with placement of an extracellular matrix to support wound healing. Although effective, this surgery can still lead to wound problems such as infection, fluid collection (seroma), wound separation (dehiscence), and delayed healing.

This study aims to compare two different solutions used to rinse the surgical wound before closing it. One solution is Irrisept, which contains 0.05% chlorhexidine gluconate, an antiseptic designed to reduce bacteria. The other is normal saline, which is the current standard rinse used in surgery. The goal is to determine whether using Irrisept can safely reduce post-operative infections and wound-related complications in patients undergoing flap closure and extracellular matrix implantation for pilonidal disease.

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) is an acquired condition involving chronic inflammation and infection in the sacrococcygeal region. Over time, PSD can lead to recurrent infections, draining tracts, abscess formation, and the need for repeated procedures. Surgical management often includes flap-based closure techniques. The bilateral gluteal fasciocutaneous flap with midline closure, combined with implantation of an extracellular matrix, is designed to provide durable coverage and improve wound healing. However, wound-related complications remain common. Reported rates of wound dehiscence for flap-based closures range from approximately 10% to 36%, and infection and seroma formation continue to be major concerns.

This prospective study evaluates whether the use of Irrisept (0.05% chlorhexidine gluconate) as an antimicrobial irrigation solution during flap closure can reduce these complications compared with standard irrigation using normal saline. The study will assess safety and effectiveness by comparing the rates of postoperative infection, seroma, hematoma, wound dehiscence, and time to complete wound healing between the two groups.

Participants will be adults undergoing bilateral gluteal fasciocutaneous flap closure with implantation of the Myriad extracellular matrix for treatment of pilonidal disease. All other aspects of surgical care will follow standard practice. Participants will be monitored after surgery for healing progress and any treatment-emergent adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent and to comply with the requirements of the Clinical Investigational Plan
2. Male or female patients aged 18 years or above
3. Patients scheduled for flap-based procedure for pilonidal disease with planned use of Irrisept or normal saline irrigation
4. Subjects who are willing and able to comply with all aspects of the treatment and evaluation schedule

Exclusion Criteria:

1. Known allergy to contents of Irrisept (chlorhexidine gluconate)
2. Full-thickness ('third degree') burns
3. Wounds with uncontrolled clinical infection (CDC Contamination Grade 4)
4. Any medical condition or serious intercurrent illness that, in the opinion of the investigator, may make it undesirable for the patient to participate in the study
5. Currently participating or has participated in another clinical study within 30 days prior to enrollment
6. Pregnant or lactating women
7. Any subject who, at the discretion of the Investigator, is not suitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events (TEAEs) | From the day of surgery through 3-month postoperative follow-up
  Proportion of participants who experience any treatment-emergent adverse event following surgery and throughout the follow-up period. Adverse events include any unfavorable or unintended sign, symptom, or medical occurrence temporally associated with the study intervention.

SECONDARY OUTCOMES:
Time to Complete Wound Healing | Up to 3 months after surgery
  Number of weeks from surgery to complete wound healing, defined as full epithelialization without drainage, dehiscence, or need for additional wound treatment.
Postoperative Infection Rate | Up to 3 months after surgery
  Proportion of participants who develop a postoperative surgical site infection, defined by clinical assessment as purulent drainage, positive wound culture, or physician diagnosis requiring antibiotics or procedural intervention.
Seroma or Hematoma Formation | Up to 3 months after surgery
  Proportion of participants who develop a postoperative seroma or hematoma confirmed by clinical exam or imaging and requiring observation or intervention.
Wound Dehiscence | Up to 3 months after surgery
  Proportion of participants who experience wound separation (partial or complete) requiring additional wound care, packing, or procedural management.

CONTACTS AND LOCATIONS:
Locations (1):
- Surgery Group LA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No